CLINICAL TRIAL: NCT02934477
Title: Prospective Assessment of Allogeneic Hematopoietic Cell Transplantation in Patients With Myelofibrosis
Status: Recruiting | Type: Observational
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Marrow Donor Program (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 16-CMS-MF; U24CA076518 (NIH)
Record Dates: First submitted 2016-09-30; First posted 2016-10-17 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis; Hematopoietic Stem Cell Transplant; Medicare
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hematopoietic Stem Cell Transplant (HCT): Patients undergoing alloHCT in a US transplant center and reported to the CIBMTR
  Interventions: Other: Hematopoietic Stem Cell Transplant
- Non-HCT: Historical non-transplant controls collected from 14 US academic centers. Centers will provide data on all consecutive patients with PMF, post-ET MF, or post-PV MF referred to their institutions between 2000 and 2012.

INTERVENTIONS:
Other: Hematopoietic Stem Cell Transplant — This observational study will compare outcomes of prospectively enrolled HCT recipients with outcomes of a cohort of age-matched non-HCT controls.
  Groups: Hematopoietic Stem Cell Transplant (HCT)

SUMMARY:
This observational study will compare outcomes of a prospectively-enrolled cohort of Hematopoietic Stem Cell Transplant (HCT) recipients with outcomes of a cohort of age-matched historical non-HCT controls. Patients undergoing alloHCT will receive HCT in a US transplant center and be reported to the Center for International Blood and Marrow Transplant Research (CIBMTR) using well-established CIBMTR report forms and data collection procedures as well as a study-specific supplemental form. Data on the historical non-HCT controls will be collected at 14 US academic centers. These centers will provide data on all consecutive patients with PMF, post-ET MF, or post-PV MF referred to their institutions between 2000 and 2012.

DETAILED DESCRIPTION:
Patients with primary MF (PMF), post-essential thrombocythemia (ET) MF, or post-polycythemia vera (PV) MF, with intermediate-2 or high-risk disease as determined by the DIPSS, and aged ≥55 at the time of DIPSS assessment are eligible for this study. For the allogeneic HCT arm of the HLA-Matched Donor HCT Study, donors must be either 6/6 HLA-matched related donors, defined by Class I (HLA-A and -B) intermediate resolution or high resolution DNA-based typing and Class II (HLA-DRBI) at high resolution DNA-based typing (but not monozygotic twins), OR an 8/8 HLA-A, -B, -C, and -DRB1 at high resolution DNA-based typing matched unrelated donors; both peripheral blood stem cells and bone marrow grafts are allowed, and all conditioning regimen intensities and graph versus host disease (GVHD) prophylaxis regimens are allowed. For the Haploidentical Donor Study, donors must be haploidentical.

This study will target accrual of 650 patients receiving alloHCT, including approximately 225 receiving myeloablative conditioning. Participating centers are expected to provide data for approximately 2,400 patients to form the non-HCT historical control cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the following criteria will be eligible for inclusion in the study:

  * PMF, post-ET MF, or post-PV MF.
  * Int-2 or high-risk disease as determined by the DIPSS.
  * Age ≥55 at the time of DIPSS assessment.
  * For the alloHCT arm:

    * Donors must be a 6/6 HLA-matched related donors, defined by Class I (HLA-A and -B) intermediate resolution or high resolution DNA-based typing and Class II (HLA-DRBI) at high resolution DNA-based typing (but not monozygotic twins) OR an 8/8 HLA-A, -B, -C, and -DRB1 at high resolution DNA-based typing matched unrelated donor identified through the National Marrow Donor Program (NMDP)/Be The Match. Donors must meet institutional or NMDP/Be The Match selection criteria; there is no age restriction for sibling donors.
    * Both peripheral blood stem cells and bone marrow grafts are allowed.
    * All conditioning regimen intensities are allowed.
    * All GVHD prophylaxis regimens are allowed.
  * Haploidentical donors are allowed in the Haploidentical Donor Study

Exclusion Criteria:

* Patients with the following criteria will be ineligible for entry into the study:

  * AlloHCT using umbilical cord blood unit(s) or HLA-mismatched adult donors (< 6/6 HLA alleles for related and < 8/8 HLA alleles for unrelated).
  * Overlap syndromes.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary MF (PMF), post-essential thrombocythemia (ET) MF, or post-polycythemia vera (PV) MF, with intermediate-2 or high-risk disease as determined by the DIPSS, and aged ≥55 at the time of DIPSS assessment are eligible for this study. For the alloHCT arm of the HLA-Matched Donor HCT Study, donors must be either 6/6 HLA-matched related donors, defined by Class I (HLA-A and -B) intermediate resolution or high resolution DNA-based typing and Class II (HLA-DRBI) at high resolution DNA-based typing (but not monozygotic twins), OR an 8/8 HLA-A, -B, -C, and -DRB1 at high resolution DNA-based typing matched unrelated donors; both peripheral blood stem cells and bone marrow grafts are allowed, and all conditioning regimen intensities and GVHD prophylaxis regimens are allowed. For the Haploidentical Donor Study, donors must be haploidentical.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2016-11; Primary Completion 2026-11 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Compare five year survival | Five years post transplant
  Compare the five-year survival probabilities from DIPSS assessment between the two study arms: alloHCT recipients (arm 1) and non-HCT therapies (ruxolitinib / best supportive care) recipients (arm 2).

SECONDARY OUTCOMES:
Compare leukemia-free survival | Five years post transplant
  Compare leukemia-free survival at five years from DIPSS assessment date to the date of progression to AML or death from any cause, whichever comes first. Two co-secondary analyses will be conducted, one for all alloHCT patients versus Arm 2 and one for the subset of patients receiving MAC prior to alloHCT versus Arm 2. Observation is censored at the date of last follow-up for patients known to be alive without leukemia. Progression to AML is defined as >20% leukemia blasts in bone marrow or in the peripheral blood.
Cumulative incidences of chronic GVHD | Five years post transplant
  Occurrence of symptoms in any organ system fulfilling the criteria of chronic GVHD. Patients are censored at last follow-up or second transplant.
Cumulative incidences of acute GVHD | Five years post transplant
  Occurrence of grade II, III, and/or IV skin, gastrointestinal, or liver abnormalities fulfilling the Consensus criteria of acute GVHD. Patients are censored at last follow-up or second transplant.
Cumulative incidence of treatment related mortality | Five years post transplant
  Death from any cause in the first 28 days post-transplantation, irrespective of relapse status. Death beyond day +28 will only be considered transplant-related if the disease is in remission. This event will be summarized as a cumulative incidence estimate with relapse/persistence as the competing risk.
The impact of certain patient, disease and HCT related factors on survival in the alloHCT arm. | Five years post transplant
  Evaluation of the impact of response to ruxolitinib therapy, patient age (<65 years vs. >= 65 years, disease duration and DIPSS on overall survival in the alloHCT arm. The time to event in the analyses will start at the time of transplant.
The impact of certain patient, disease and HCT related factors on leukemia free survival in the alloHCT arm. | Five years post transplant
  Evaluation of the impact of response to ruxolitinib therapy, patient age (<65 vs. >= 65 years), disease duration and DIPSS on leukemia free survival in the alloHCT arm. The time to event in the analyses will start at the time of transplant.
The impact of certain patient, disease and HCT related factors on hematopoietic recovery in the alloHCT arm. | Five years post transplant
  Evaluation of the impact of response to ruxolitinib therapy, patient age (<65 vs >=65 years), disease duration and DIPSS on hematopoietic recovery in the alloHCT arm. The time to event in the analyses will start at the time of transplant.
The impact of certain patient, disease and HCT related factors on acute and chronic GVHD in the alloHCT arm. | Five years post transplant
  Evaluation of the impact of response to ruxolitinib therapy, patient age (<65 vs >= 65 years), disease duration and DIPSS on acute and chronic GVHD in the alloHCT arm. The time to event in the analyses will start at the time of transplant.
The impact of certain patient, disease and HCT related factors on treatment related mortality in the alloHCT arm. | Five years post transplant.
  Evaluation of the impact of response to ruxolitinib therapy, patient age (<65 vs >=65 years), disease duration, and DIPSS on treatment related mortality in the alloHCT arm. The time to event in the analyses will start at the time of transplant.
The impact of certain patient, disease and HCT related factors on relapse. | Five years post transplant.
  Evaluation of the impact of response to ruxolitinib therapy, patient age (65 vs >=65 years), disease duration and DIPSS on relapse in the alloHCT arm. The time to event in the analyses will start at the time of transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Wael Saber, MD, Study Chair — Medical College of Wisconsin; Laura Michaelis, MD, Study Chair — Medical College of Wisconsin
Locations (1):
- Center for International Blood and Marrow Transplant Research, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: CIBMTR — https://www.cibmtr.org/pages/index.aspx